CLINICAL TRIAL: NCT00207324
Title: A Phase III Study of the Efficacy of Silver Leaf Nylon Dressing in the Prevention of Severe Skin Reactions in the Inframammary Skin Fold of Patients Receiving Adjuvant Whole Breast Radiotherapy
Brief Title: The Use of Silver Leaf Dressing in the Prevention of Radiotherapy Induced Skin Reactions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: R03-0030
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Silver Leaf Dressing

SUMMARY:
The hypothesis is that silver leaf nylon dressing reduces the percentage of patients developing brisk erythema and moist desquamation while undergoing whole breast radiotherapy. The secondary hypothesis is that silver leaf nylon dressing reduces breast-related symptoms of pain, itching and burning sensation in patients receiving whole breast radiotherapy.

DETAILED DESCRIPTION:
Purpose: The delivery of whole breast radiotherapy to women with a deep inframammary fold frequently results in a marked skin reaction (brisk erythema and/or moist desquamation). The main aim of this study is to compare the efficacy of prophylactic silver leaf nylon dressings with standard skin care against standard skin care alone in the prevention of brisk erythema and moist desquamation. A secondary aim of the study is to assess whether the use of silver leaf nylon dressings can reduce breast-related symptoms of pain, burning sensation and itching in women undergoing whole breast radiotherapy.

Hypothesis: The hypothesis is that silver leaf nylon dressing reduces the percentage of patients developing brisk erythema and moist desquamation while undergoing whole breast radiotherapy. The secondary hypothesis is that silver leaf nylon dressing reduces breast-related symptoms of pain, itching and burning sensation in patients receiving whole breast radiotherapy. The null hypotheses are that there is no reduction in brisk erythema, moist desquamation or breast-related symptoms in patients undergoing whole breast radiotherapy with the use of silver leaf nylon dressing.

Justification: Severe skin reactions are common in patients with a deep inframammary fold who undergo whole breast radiotherapy. It may be possible to reduce the severity of skin reactions in this population of patients with the use of silver leaf nylon dressing. This might make whole breast radiotherapy more tolerable for patients.

Objectives: The objectives of this study are to compare the severity of skin reactions of patients with a deep inframammary skin fold undergoing whole breast radiotherapy (using the Radiation Therapy Oncology Group scoring system, as well as a supplementary scoring system) between the experimental arm and the control arm, and to compare the severity of breast- related symptoms (using visual analogue scales), topical steroid use and analgesic use between the two study arms.

Research Method: This will be a single blind randomised controlled trial. The target population comprises patients with a deep inframammary fold undergoing whole breast radiotherapy. Patients will be randomised to follow standard skin care recommendations throughout radiotherapy treatment (control arm) or to follow these recommendations in addition to using a silver leaf nylon dressing (experimental arm). Randomisation will be stratified for the delivery of prior chemotherapy and for the radiotherapy fractionation schedule (extended versus standard).

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with completely excised stage I or II invasive breast cancer, or DCIS, who have undergone breast-conserving surgery and are scheduled to undergo adjuvant breast radiotherapy will be eligible for this study if they are at increased risk of radiodermatitis at the inframammary fold due to breast size or shape (i.e at least 2cm of skin apposition at the inframammary fold, and/or brassiere cup size C or greater).
2. Patients undergoing nodal radiotherapy are eligible if criterion 1 is met
3. Patients undergoing boost radiotherapy are eligible if criterion 1 is met, but only if the boost volume does not include any part of the breast inferior to the nipple line
4. Patients may be entered into other local or national trials unless these involve an alteration to standard skin care or altered breast radiotherapy technique

Exclusion Criteria:

* inability to give informed consent
* inability to comply with experimental arm of trial
* failure of healing of the surgical scar or significant post-operative infection of the wound
* prior radiotherapy to either breast or to the chest
* presence of significant connective tissue disease (e.g. systemic sclerosis, systemic lupus erythematosis)
* known radiation hypersensitivity phenotype (e.g. ataxia telangiectasia etc)
* inability to return for assessment at one week following completion of radiotherapy
* allergy to silver

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
silver leaf nylon dressing reduces the percentage of patients developing brisk erythema and moist desquamation while undergoing whole breast radiotherapy

SECONDARY OUTCOMES:
silver leaf nylon dressing reduces breast-related symptoms of pain, itching and burning sensation in patients receiving whole breast radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Christina Parsons, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada